CLINICAL TRIAL: NCT05499923
Title: Quantitative Measurement of the Adhesive Remnant Index Using Two Different Debonding Techniques: A Split-mouth Randomized Clinical Trial
Brief Title: Quantitative Measurement of ARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Lahore Medical College and Institute of Dentistry (Other)
Responsible Party: Principal Investigator, Haris Khan, Professor, CMH Lahore Medical College and Institute of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERC/CMH/LMC/621
Record Dates: First submitted 2022-06-21; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Orthodontic Appliance Complication
Keywords: Bracket Debonding , Wing method, Base method , ARI
MeSH Terms: interventions — Dental Debonding

STUDY DESIGN:
Intervention Model Description: Split mouth design
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients were blinded for the technique used in each quadrant and also the outcome assessors were blinded about the technique used for debonding brackets.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wing method of debonding (Active Comparator): In this method after removal of the orthodontic wire, each bracket would be gripped mesiodistally by a conventional bracket debonding plier at the level of wings and a squeezing force would be applied.
  Interventions: Device: Debonding
- Base method of debonding (Active Comparator): In this method after removal of the orthodontic wire, each bracket would be gripped mesiodistally by a conventional bracket debonding plier at the level of the bracket base and a squeezing force would be applied.
  Interventions: Device: Debonding

INTERVENTIONS:
Device: Debonding — Debonding of orthodontic brackets with wing or base method with a conventional debonding plier

SUMMARY:
A crucial step at end of debonding is to evaluate the site of bond failure. An accurate assessment of the site of bond failure will allow the clinician to select an optimum method for adhesive remnant removal from the enamel surface.

The aim of this study is to do a randomized clinical trial to measure adhesive remanent index quantitively after debonding with wing and base method of debonding

DETAILED DESCRIPTION:
After informed consent data would be collected from patients who are undergoing debonding of orthodontic brackets after comprehensive orthodontic treatment of at least 2 years. Only the cases which have no loose anterior upper and lower brackets for the last 6 months would be randomly allocated to one of the two sides in each arch for debonding with a specific technique. A protocol of block randomization would be followed for this study. Debonding of brackets would be done either by wing or base method in a split fashion after removal of orthodontic wires. The patient would be explained that both methods are conventional used and are safe for debonding. After debonding each bracket the patient would be asked for the level of pain he felt during the debonding of that specific bracket. The patient will explain the pain level on a scale of 0-10 with 0 referring to no pain while 10 referring to maximum pain. After debonding a digital microscope (Supereyes) would be used along with plastic tubing for taking the adhesive remanent pictures intraorally from the labial surface of teeth. The plastic tubing would have a calibrated scale attached to it. For each new patient, a new tubing or disinfected tubing would be used. The available data would be measured extra orally on a computer-based software (ImageJ). Variable like age, gender, oral hygiene, ARI, side of adhesive flush, and pain would be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* All the patients undergoing comprehensive orthodontic treatment by fixed orthodontics
* No reporting of bracket failure in the last 6 months.
* Same company metal brackets used.
* Same adhesive used with same bonding protcol

Exclusion Criteria:

* Syndromic patient
* An episode of bracket failure in the last six months
* Short-term orthodontic treatment

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 148 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Adhesive remnant index | 6 months
  Quantitative Measurement of adhesive remnant index by a digital handheld microscope

SECONDARY OUTCOMES:
Patient reported outcome: Pain | 6 months
  After debonding each bracket patient will score the pain level on a scale of 0-10 with 0 referring to no pain while 10 referring to maximum pain

OTHER OUTCOMES:
Assessor reported outcomes | 6 months
  Corrosion on labial surface of teeth and flush of adhesive noticed by the clinician by visual inspection and reported by yes or no

CONTACTS AND LOCATIONS:
Locations (1):
- Haris Khan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No